CLINICAL TRIAL: NCT01550315
Title: A Pilot Study of the Effect of Dietary Sodium Intake on Assessments of Vascular Endothelium
Brief Title: Effect of Dietary Sodium Intake on Vascular Endothelium
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Alfredo Gamboa, Research Associate Professor of Medicine, Vanderbilt University Medical Center
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 111577; R01HL102387 (NIH)
Record Dates: First submitted 2012-03-02; First posted 2012-03-09 (Estimated); Results first posted 2022-01-05 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2021-12

CONDITIONS: Postural Tachycardia Syndrome (POTS)
Keywords: POTS; endothelial function; high salt vs low salt diet; PAT protocol; Calf blood flow; forearm mediated dilation
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome | interventions — Clinical Protocols; Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Sodium - POTS & Controls (Active Comparator): Subjects will receive a high sodium diet for 4-5 days prior to study day. Procedures include: blood work, urine collection, Pulsitile Arterial Tonometry (PAT), PAT analysis, Calf Blood Flow in Reactive Hyperemia (CBF-RH), & evaluation of forearm-mediated dilation.
  Interventions: Procedure: Pulsitile Arterial Tonometry (PAT) Protocol; Device: Calf Blood Flow in Reactive Hyperemia (CBF-RH); Device: Evaluation of Forearm-Mediated Dilation
- Low Sodium Diet (POTS & Controls) (Other): Participants will consume a very low sodium diet (10 mEq/day) for 4-5 days prior to study day.
  Procedures include: blood work, urine collection, Pulsitile Arterial Tonometry (PAT), PAT analysis, Calf Blood Flow in Reactive Hyperemia (CBF-RH), & evaluation of forearm-mediated dilation.
  Interventions: Procedure: Pulsitile Arterial Tonometry (PAT) Protocol; Device: Calf Blood Flow in Reactive Hyperemia (CBF-RH); Device: Evaluation of Forearm-Mediated Dilation

INTERVENTIONS:
Procedure: Pulsitile Arterial Tonometry (PAT) Protocol — * A blood pressure cuff will be placed on one upper arm (study arm; non-dominant), while the contralateral arm will serve as a control (control arm).
  * RH-PAT probes will be placed on one finger (finger II, III, or IV) of each hand (same finger on both hands). The fingers on either side of the one with the probe will be separated using soft sponge rings.
  * Continuous recording of pulsatile blood volume responses from both hands will be initiated.
  * After a 10-min equilibration period, the blood pressure cuff on the study arm will be inflated to 60 mm Hg above systolic pressure for 5 min. The cuff will then be deflated to induce reactive hyperemia, PAT recording will be stopped.
  Other Names: EndoPat
Device: Calf Blood Flow in Reactive Hyperemia (CBF-RH) — Calf blood flow (CBF) will be determined using venous occlusion plethysmography and calibrated mercury strain-gauges during reactive hyperemia after a 5 min of ischemia of the distal limb. Strain-gauges will be applied to the widest part of the non-dominant calf (~10 cm below patella). Participants will remain quietly supine for 10 min with legs elevated on foam pads above the right atrium to achieve stable baseline measurements of CBF. The venous occlusion cuff is inflated for 4 seconds at 8 seconds intervals, while monitoring the change in resistance in the system, pressure inside the measuring cuff, and 5-10 determinations are performed
  Other Names: Hokansan strain guage venous plethysmography
Device: Evaluation of Forearm-Mediated Dilation — The arm will be kept extended and immobilized at heart level. Brachial artery diameter will be measured using a high resolution ultrasonography using a linear array probe with a 5 to 17 MHz frequency range. The brachial artery will be imaged in longitudinal sections, 5-10 cm proximal to placement of an occlusion cuff in the dominant forearm just below the antecubital fossa. The probe will be held with a stereotaxic holder with micrometer movement capabilities.
  Other Names: Ultrasound

SUMMARY:
The investigators will test the hypothesis that markers of vascular endothelial dysfunction will be exaggerated acutely with an extreme high sodium diet compared to an extreme low-sodium diet. The investigators will compare patients with postural orthostatic tachycardia (POTS) to healthy control subjects.

DETAILED DESCRIPTION:
The study will involve a crossover design in which each subject will be assessed (as below) while on a very low-sodium (10 mEq/day) diet compared with a very high-sodium diet. These acute dietary interventions will be part of the parent study ("Dietary Salt in Postural Tachcyardia Syndrome" funded by R01 HL102387) for 4-5 days at the time of the study. Dietary success will be assessed using a 24h urine for sodium and creatinine as a part of the parent study.

Blood will be drawn and collected in a fasting state for future assay and analysis of the following tests:

* Glucose, Insulin (glucose impairment, insulin resistance)
* Fasting lipid profile
* C-Reactive Protein (hsCRP) (inflammatory state)
* Inflammatory cytokines (inflammatory state)
* aliquots (future analysis)

Pulsitile Arterial Tonometry (PAT) Protocol Calf Blood Flow in Reactive Hyperemia (CBF-RH) - venous occlusion plethysmography Evaluation of Forearm-Mediated Dilation

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be enrolled in the parent study "Dietary Salt in Postural Tachcyardia Syndrome" funded by R01 HL102387 Postural Tachycardia Syndrome
* Diagnosed with postural tachycardia syndrome by the Vanderbilt Autonomic Dysfunction Center
* Subjects will be enrolled in the parent study "Dietary Salt in Postural Tachcyardia Syndrome" funded by R01 HL102387
* Postural Tachycardia Syndrome
* Diagnosed with postural tachycardia syndrome by the Vanderbilt Autonomic Dysfunction Center
* Increase in heart rate ≥30 beats/min with position change from supine to standing (10 minutes)
* Chronic symptoms consistent with POTS that are worse when upright and get better with recumbence Control Subjects
* Healthy, non-obese, non-smokers without orthostatic tachycardia
* Selected to match profiles of POTS patients (gender, age)
* Not using vasoactive medication
* Age between 18-60 years
* Male and female subjects are eligible.
* Able and willing to provide informed consent

Exclusion Criteria:

* Overt cause for postural tachycardia (such as acute dehydration)
* Inability to give, or withdrawal of, informed consent
* Pregnant
* Other factors which in the investigator's opinion would prevent the subject from completing the protocol.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2012-04; Primary Completion 2020-12 (Actual); Study Completion 2021-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Satish R Raj, MD MSCI, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Background] Clarkson P, Celermajer DS, Powe AJ, Donald AE, Henry RM, Deanfield JE. Endothelium-dependent dilatation is impaired in young healthy subjects with a family history of premature coronary disease. Circulation. 1997 Nov 18;96(10):3378-83. doi: 10.1161/01.cir.96.10.3378. PMID 9396430
- [Background] Al Suwaidi J, Higano ST, Holmes DR Jr, Lennon R, Lerman A. Obesity is independently associated with coronary endothelial dysfunction in patients with normal or mildly diseased coronary arteries. J Am Coll Cardiol. 2001 May;37(6):1523-8. doi: 10.1016/s0735-1097(01)01212-8. PMID 11345360
- [Background] Boger RH, Bode-Boger SM, Szuba A, Tsao PS, Chan JR, Tangphao O, Blaschke TF, Cooke JP. Asymmetric dimethylarginine (ADMA): a novel risk factor for endothelial dysfunction: its role in hypercholesterolemia. Circulation. 1998 Nov 3;98(18):1842-7. doi: 10.1161/01.cir.98.18.1842. PMID 9799202
- [Background] Mangin EL Jr, Kugiyama K, Nguy JH, Kerns SA, Henry PD. Effects of lysolipids and oxidatively modified low density lipoprotein on endothelium-dependent relaxation of rabbit aorta. Circ Res. 1993 Jan;72(1):161-6. doi: 10.1161/01.res.72.1.161. PMID 8417838
- [Background] Vergnani L, Hatrik S, Ricci F, Passaro A, Manzoli N, Zuliani G, Brovkovych V, Fellin R, Malinski T. Effect of native and oxidized low-density lipoprotein on endothelial nitric oxide and superoxide production : key role of L-arginine availability. Circulation. 2000 Mar 21;101(11):1261-6. doi: 10.1161/01.cir.101.11.1261. PMID 10725285
- [Background] Landmesser U, Merten R, Spiekermann S, Buttner K, Drexler H, Hornig B. Vascular extracellular superoxide dismutase activity in patients with coronary artery disease: relation to endothelium-dependent vasodilation. Circulation. 2000 May 16;101(19):2264-70. doi: 10.1161/01.cir.101.19.2264. PMID 10811593
- [Background] Quyyumi AA, Dakak N, Andrews NP, Husain S, Arora S, Gilligan DM, Panza JA, Cannon RO 3rd. Nitric oxide activity in the human coronary circulation. Impact of risk factors for coronary atherosclerosis. J Clin Invest. 1995 Apr;95(4):1747-55. doi: 10.1172/JCI117852. PMID 7706483
- [Background] Appel LJ, Frohlich ED, Hall JE, Pearson TA, Sacco RL, Seals DR, Sacks FM, Smith SC Jr, Vafiadis DK, Van Horn LV. The importance of population-wide sodium reduction as a means to prevent cardiovascular disease and stroke: a call to action from the American Heart Association. Circulation. 2011 Mar 15;123(10):1138-43. doi: 10.1161/CIR.0b013e31820d0793. Epub 2011 Jan 13. No abstract available. PMID 21233236
- [Background] Meneton P, Jeunemaitre X, de Wardener HE, MacGregor GA. Links between dietary salt intake, renal salt handling, blood pressure, and cardiovascular diseases. Physiol Rev. 2005 Apr;85(2):679-715. doi: 10.1152/physrev.00056.2003. PMID 15788708
- [Background] MENEELY GR, BALL CO. Experimental epidemiology of chronic sodium chloride toxicity and the protective effect of potassium chloride. Am J Med. 1958 Nov;25(5):713-25. doi: 10.1016/0002-9343(58)90009-3. No abstract available. PMID 13582981
- [Background] Strazzullo P, D'Elia L, Kandala NB, Cappuccio FP. Salt intake, stroke, and cardiovascular disease: meta-analysis of prospective studies. BMJ. 2009 Nov 24;339:b4567. doi: 10.1136/bmj.b4567. PMID 19934192
- [Background] Dishy V, Sofowora GG, Imamura H, Nishimi Y, Xie HG, Wood AJ, Stein CM. Nitric oxide production decreases after salt loading but is not related to blood pressure changes or nitric oxide-mediated vascular responses. J Hypertens. 2003 Jan;21(1):153-7. doi: 10.1097/00004872-200301000-00025. PMID 12544447
- [Background] Fujiwara N, Osanai T, Kamada T, Katoh T, Takahashi K, Okumura K. Study on the relationship between plasma nitrite and nitrate level and salt sensitivity in human hypertension : modulation of nitric oxide synthesis by salt intake. Circulation. 2000 Feb 29;101(8):856-61. doi: 10.1161/01.cir.101.8.856. PMID 10694524
- [Background] Kuvin JT, Patel AR, Sliney KA, Pandian NG, Sheffy J, Schnall RP, Karas RH, Udelson JE. Assessment of peripheral vascular endothelial function with finger arterial pulse wave amplitude. Am Heart J. 2003 Jul;146(1):168-74. doi: 10.1016/S0002-8703(03)00094-2. PMID 12851627
- [Background] Rozanski A, Qureshi E, Bauman M, Reed G, Pillar G, Diamond GA. Peripheral arterial responses to treadmill exercise among healthy subjects and atherosclerotic patients. Circulation. 2001 Apr 24;103(16):2084-9. doi: 10.1161/01.cir.103.16.2084. PMID 11319199
- [Background] Meredith IT, Currie KE, Anderson TJ, Roddy MA, Ganz P, Creager MA. Postischemic vasodilation in human forearm is dependent on endothelium-derived nitric oxide. Am J Physiol. 1996 Apr;270(4 Pt 2):H1435-40. doi: 10.1152/ajpheart.1996.270.4.H1435. PMID 8967386
- [Background] Dakak N, Husain S, Mulcahy D, Andrews NP, Panza JA, Waclawiw M, Schenke W, Quyyumi AA. Contribution of nitric oxide to reactive hyperemia: impact of endothelial dysfunction. Hypertension. 1998 Jul;32(1):9-15. doi: 10.1161/01.hyp.32.1.9. PMID 9674631
- [Background] Higashi Y, Sasaki S, Nakagawa K, Matsuura H, Kajiyama G, Oshima T. A noninvasive measurement of reactive hyperemia that can be used to assess resistance artery endothelial function in humans. Am J Cardiol. 2001 Jan 1;87(1):121-5, A9. doi: 10.1016/s0002-9149(00)01288-1. PMID 11137850
- [Background] Wilkinson IB, Qasem A, McEniery CM, Webb DJ, Avolio AP, Cockcroft JR. Nitric oxide regulates local arterial distensibility in vivo. Circulation. 2002 Jan 15;105(2):213-7. doi: 10.1161/hc0202.101970. PMID 11790703
- [Background] Noon JP, Haynes WG, Webb DJ, Shore AC. Local inhibition of nitric oxide generation in man reduces blood flow in finger pulp but not in hand dorsum skin. J Physiol. 1996 Jan 15;490 ( Pt 2)(Pt 2):501-8. doi: 10.1113/jphysiol.1996.sp021161. PMID 8821146
- [Background] Nohria A, Gerhard-Herman M, Creager MA, Hurley S, Mitra D, Ganz P. Role of nitric oxide in the regulation of digital pulse volume amplitude in humans. J Appl Physiol (1985). 2006 Aug;101(2):545-8. doi: 10.1152/japplphysiol.01285.2005. Epub 2006 Apr 13. PMID 16614356
- [Background] Thijssen DH, Black MA, Pyke KE, Padilla J, Atkinson G, Harris RA, Parker B, Widlansky ME, Tschakovsky ME, Green DJ. Assessment of flow-mediated dilation in humans: a methodological and physiological guideline. Am J Physiol Heart Circ Physiol. 2011 Jan;300(1):H2-12. doi: 10.1152/ajpheart.00471.2010. Epub 2010 Oct 15. PMID 20952670
- [Background] Deanfield J, Donald A, Ferri C, Giannattasio C, Halcox J, Halligan S, Lerman A, Mancia G, Oliver JJ, Pessina AC, Rizzoni D, Rossi GP, Salvetti A, Schiffrin EL, Taddei S, Webb DJ; Working Group on Endothelin and Endothelial Factors of the European Society of Hypertension. Endothelial function and dysfunction. Part I: Methodological issues for assessment in the different vascular beds: a statement by the Working Group on Endothelin and Endothelial Factors of the European Society of Hypertension. J Hypertens. 2005 Jan;23(1):7-17. doi: 10.1097/00004872-200501000-00004. PMID 15643116
- [Background] Bonetti PO, Pumper GM, Higano ST, Holmes DR Jr, Kuvin JT, Lerman A. Noninvasive identification of patients with early coronary atherosclerosis by assessment of digital reactive hyperemia. J Am Coll Cardiol. 2004 Dec 7;44(11):2137-41. doi: 10.1016/j.jacc.2004.08.062. PMID 15582310
- [Background] Centers for Disease Control and Prevention (CDC). Vital signs: prevalence, treatment, and control of hypertension--United States, 1999-2002 and 2005-2008. MMWR Morb Mortal Wkly Rep. 2011 Feb 4;60(4):103-8. PMID 21293325
- [Derived] Smith EC, Celedonio J, Nwazue VC, Garland EM, Paranjape SY, Chopoorian AH, Wahba A, Biaggioni I, Black B, Shibao CA, Diedrich A, Okamoto LE, Raj SR, Gamboa A. High-sodium diet does not worsen endothelial function in female patients with postural tachycardia syndrome. Clin Auton Res. 2021 Aug;31(4):563-571. doi: 10.1007/s10286-021-00772-y. Epub 2021 Mar 10. PMID 33689063

RESULTS

PARTICIPANT FLOW:
Groups:
- High Sodium First- POTS: POTS patients received a high salt diet (300 mEq/day) for 6 days in a randomized crossover design and two weeks after, were crossover to receive a low high diet for 6 days
- Low Sodium Diet First-POTS: POTS patients received a low salt diet (10 mEq/day) for 6 days in a randomized crossover design, and two weeks later received a high salt diet.
- High Sodium First- Controls: Healthy Controls received a high salt diet (300 mEq/day) for 6 days in a randomized crossover design and two weeks after, received a low high diet for 6 days
- Low Sodium First-Controls: Healthy Controls received a low salt diet (10 mEq/day) for 6 days in a randomized crossover design, and two weeks later received a high salt diet.
Period: Overall Study
Arm/Group | High Sodium First- POTS | Low Sodium Diet First-POTS | High Sodium First- Controls | Low Sodium First-Controls
Started | 7 | 7 | 6 | 7
Completed | 7 | 7 | 6 | 7
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study POTS: POTS patients received high sodium diet for 4-5 days prior to study day. Then received either a high sodium diet (300 mEq/day) diet for 6 days, then after 2 weeks were randomized in a crossover design to receive a low sodium diet (10 mEq/day) diet for 6 days, or viceversa (first low then high salt diet). All POTS patients received both diets.
  Evaluation of Forearm-Mediated Dilation: The arm will be kept extended and immobilized at heart level. Brachial artery diameter will be measured using a high resolution ultrasonography using a linear array probe with a 5 to 17 MHz frequency range. The brachial artery will be imaged in longitudinal sections, 5-10 cm proximal to placement of an occlusion cuff in the dominant forearm just below the antecubital fossa. The probe will be held with a stereotaxic holder with micrometer movement capabilities.
- All Study Controls: Healthy controls received high sodium diet for 4-5 days prior to study day. Then received either a high sodium diet (300 mEq/day) diet for 6 days, then after 2 weeks were randomized in a crossover design to receive a low sodium diet (10 mEq/day) diet for 6 days, or viceversa (first low then high salt diet). All healthy controls received both diets.
  Evaluation of Forearm-Mediated Dilation: The arm will be kept extended and immobilized at heart level. Brachial artery diameter will be measured using a high resolution ultrasonography using a linear array probe with a 5 to 17 MHz frequency range. The brachial artery will be imaged in longitudinal sections, 5-10 cm proximal to placement of an occlusion cuff in the dominant forearm just below the antecubital fossa. The probe will be held with a stereotaxic holder with micrometer movement capabilities.
- Total: Total of all reporting groups
Arm/Group | All Study POTS | All Study Controls | Total
Number analyzed (Participants) | 14 | 13 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 35 (8) | 31 (6) | 33 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 27
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 00 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 14 | 13 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 13 | 27

OUTCOME MEASURES:

1. Primary Outcome: FMD (% Change)
Description: The primary analysis will involve a non-parametric, paired, Signed Rank test of flow mediated dilation (FMD) between all subjects (POTS & control subjects) on the high sodium diet vs low sodium diet
Time Frame: FMD was assessed on the morning of day 7, after 6 days of being on either a high salt diet or a low salt diet.
Measure: Mean (Standard Deviation); unit: percentage of change
Groups:
- High Sodium POTS: POTS patients received a high sodium diet for 4-5 days prior to study day. After enrollment, they received a high salt diet (300 mEq/day) diet for 6 days in a randomized crossover design.
  Evaluation of Forearm-Mediated Dilation: The arm will be kept extended and immobilized at heart level. Brachial artery diameter will be measured using a high resolution ultrasonography using a linear array probe with a 5 to 17 MHz frequency range. The brachial artery will be imaged in longitudinal sections, 5-10 cm proximal to placement of an occlusion cuff in the dominant forearm just below the antecubital fossa. The probe will be held with a stereotaxic holder with micrometer movement capabilities.
- Low Sodium Diet POTS: POTS patients received a high sodium diet for 4-5 days prior to study day. After enrollment, they received either a low-sodium (LS; 10 mEq/day) diet for 6 days.
  Evaluation of Forearm-Mediated Dilation: The arm will be kept extended and immobilized at heart level. Brachial artery diameter will be measured using a high resolution ultrasonography using a linear array probe with a 5 to 17 MHz frequency range. The brachial artery will be imaged in longitudinal sections, 5-10 cm proximal to placement of an occlusion cuff in the dominant forearm just below the antecubital fossa. The probe will be held with a stereotaxic holder with micrometer movement capabilities.
- High Sodium Controls: Healthy controls received a high sodium diet for 4-5 days prior to study day. After enrollment, they received a high salt diet (300 mEq/day) diet for 6 days in a randomized crossover design.
  Evaluation of Forearm-Mediated Dilation: The arm will be kept extended and immobilized at heart level. Brachial artery diameter will be measured using a high resolution ultrasonography using a linear array probe with a 5 to 17 MHz frequency range. The brachial artery will be imaged in longitudinal sections, 5-10 cm proximal to placement of an occlusion cuff in the dominant forearm just below the antecubital fossa. The probe will be held with a stereotaxic holder with micrometer movement capabilities.
- Low Sodium Controls: Healthy controls received a high sodium diet for 4-5 days prior to study day. After enrollment, they received either a low-sodium (LS; 10 mEq/day) diet for 6 days.
  Evaluation of Forearm-Mediated Dilation: The arm will be kept extended and immobilized at heart level. Brachial artery diameter will be measured using a high resolution ultrasonography using a linear array probe with a 5 to 17 MHz frequency range. The brachial artery will be imaged in longitudinal sections, 5-10 cm proximal to placement of an occlusion cuff in the dominant forearm just below the antecubital fossa. The probe will be held with a stereotaxic holder with micrometer movement capabilities.
Arm/Group | High Sodium POTS | Low Sodium Diet POTS | High Sodium Controls | Low Sodium Controls
Number analyzed (Participants) | 14 | 14 | 13 | 13
percentage of change | 12.75 (43.77) | 11.65 (4.93) | 11.43 (4.26) | 12.75 (4.49)

ADVERSE EVENTS:
Time Frame: Adverse events were collected while the participants were receiving the study diets. For all participants (POTS and Controls), it involved at least 22 days: 4 days prior to randomization, 6 days in the first diet, the first study day, 2 weeks of washout, 6 days in the second diet, and the last study day.
Groups:
- High Sodium - POTS: POTS patients received a high salt diet (300 mEq/day) for 6 days in a randomized crossover design
- Low Sodium Diet - POTS: POTS patients received a low salt diet (10 mEq/day) for 6 days in a randomized crossover design
- High Sodium - Controls: Healthy controls received a high salt diet (300 mEq/day) for 6 days in a randomized crossover design
- Low Sodium - Controls: Healthy controls received a low salt diet (10 mEq/day) for 6 days in a randomized crossover design
Arm/Group | High Sodium - POTS | Low Sodium Diet - POTS | High Sodium - Controls | Low Sodium - Controls
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14 | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/13 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2014-05-28): https://cdn.clinicaltrials.gov/large-docs/15/NCT01550315/Prot_SAP_ICF_000.pdf